CLINICAL TRIAL: NCT04421898
Title: 3D Modelling and Morphometric Characterisation of the Skull Deformations in Congenital Muscular Torticollis : Development of Physiopathological Sequences
Brief Title: 3D Characterisation of the Skull Base Deformation in Congenital Muscular Torticollis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: EA2415 - Montpellier University, Montpellier, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0303
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Congenital Torticollis; Positionnel Skull Deformation
Keywords: Skull base; Petrous Bone; Plagiocephaly; Congenital Muscular Torticollis; Sternocleidomastoid muscle; Craniovertebral junction
MeSH Terms: conditions — Congenital torticollis; Plagiocephaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: group 1 : infants with congenital muscular torticollis
- group 2: group 2 : healthy , without congenital muscular torticollis

SUMMARY:
The congenital muscular torticollis (CMT) is defined by an abnormal posture of the head and the neck compared to shoulders' level of the newborn. The mainly affected muscle is the sternocleidomastoid muscle (SCM) causing a lateral inclination of the head on the side affected by the CMT and a rotation on the opposite side. CMT comes with asymmetricalndeformation of the skull or plagiocephaly, facial asymmetry, skull and cranio-vertebral deformatioes in CMT are the results of a complex mechanism of biomechanical stresses upon a developing skull. The hypothesis of a traction force on the base of the skull from the SCM could explain most of all the asymmetrical deformatios encountered in CMT. It would be associated to a compression force at the occipital level

DETAILED DESCRIPTION:
The congenital muscular torticollis (CMT) is defined by an abnormal posture of the head and the neck compared to shoulders' level of the newborn. The mainly affected muscle is the sternocleidomastoid muscle (SCM) causing a lateral inclination of the head on the side affected by the CMT and a rotation on the opposite side. It is the third cause of neonatal deformation and affect nearly one newborn out of six, most of the time transiently.

Three types of CMT exist : CMT secondary to a tonus disorder (postural torticollis), CMT presenting a tumor on the SCM and CMT caused by a retraction and fibrosis of the SCM.

The exact aetiology of CMT is not well known. However, per partum intrauterine restrictive stress is very much involved in the genesis of CMT.Treatment is mainly based on physiotherapy, it needs to be started early and associated with parental education. In the event of a failure of the physical therapy, a surgical treatment can be considered. CMT is a risk factor for delayed psychomotor development and can lead to long term sequelae in motor coordination.

CMT comes with asymmetrical deformation of the skull or plagiocephaly. Skull deformation in plagiocephaly is a 3D deformation affecting the calvaria, the skull base and the face. The skull base asymmetry can be found at the mastoid process of the petrous bone, insertion of the SCM on the base of the skull. The facial asymmetry in CMT can have an aesthetic impact on the face or a functional impact on the long term occlusion. CMT also come with abnormalities of the junction between the skull and the vertebrae, they impact the cervical mobility and foster premature arthrosis. The CMT care will modify the seriousness of the skull and face deformation, severity is major in neglected or not treated CMT.

Plagiocephly, facial asymmetry, skull and cranio-vertebral deformation in CMT are the results of a complex mechanism of biomechanical stresses upon a developing skull. These stresses appear in a context of intrauterine postural distortions and/or during postnatal distorting sequences. The SCM responsible for CMT is inserted on the mastoid process of the petrous bone for its base of the skull insertion, the petrous bone is a fundamental component in the biomechanics of the base of the skull.

The hypothesis of a traction force on the base of the skull from the SCM could explain most of all the 3D asymmetrical deformation encountered in CMT. It would be associated to a compression force at the occipital level particularly linked to a sleep position of the infants on their back, position that is now recommended.

The traction force is different depending on the CMT with no or little force in postural torticollis and strong and constant forces in torticollis with fibrosis.

ELIGIBILITY:
Inclusion criteria:

* subjects with CMT and skull deformation referenced in Data base images of CT scan

Exclusion criteria:

- incomplete clinical or CT-scan data

Max Age: 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pathologic group : children with CMT and skull deformation Control group: healthy subject from 0 to 36 month without CMT or skull deformation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
create a physiopathological 3D model of skull deformation for each type of CMTs) | 1 day
  create a physiopathological 3D model of skull deformation for each type of CMTs)

SECONDARY OUTCOMES:
Characterisation of the skull base asymmetry and cranioverterbral deformation | 1 day
  Characterisation of the skull base asymmetry and cranioverterbral deformation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CAPTIER, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC